CLINICAL TRIAL: NCT04396899
Title: Safety and Efficacy of Induced Pluripotent Stem Cell-derived Engineered Human Myocardium as Biological Ventricular Assist Tissue in Terminal Heart Failure
Acronym: BioVAT-HF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); University Medical Center Freiburg (Other); Repairon GmbH (Unknown)
Responsible Party: Principal Investigator, Karsten Gavenis, on behalf of Principal Investigator Prof. Seidler and Study Director Prof. Zimmermann, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02289
Record Dates: First submitted 2020-05-11; First posted 2020-05-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EHM Implantation (Other): All patients will receive EHM implant
  Interventions: Biological: EHM implantation

INTERVENTIONS:
Biological: EHM implantation — Implantation of EHM on dysfunctional left or right ventricular myocardium in patients with HFrEF (EF <35%).

SUMMARY:
The BioVAT-HF trial will test the hypothesis that cardiomyocyte implantation via engineered heart muscle (EHM), the proposed investigational medicinal product (IMP; designated "Biological Ventricular Assist Tissue" or BioVAT), results in sustainable remuscularization and biological enhancement of myocardial performance in the failing heart. EHM are constructed from defined mixtures of induced pluripotent stem cell (iPSC)-derived cardiomyocytes and stromal cells in a bovine collagen type I hydrogel. Comprehensive preclinical testing confirmed the rationale for the clinical translation of the myocardial remuscularization strategy by EHM implantation. The patient target population for EHM therapy is patients suffering from advanced heart failure with reduced ejection fraction (HFrEF; EF: ≤35%) and no realistic option for heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. HFrEF (EF ≤ 35%) as assessed by high-resolution echocardiography or MRI
2. No realistic chance or not eligible for heart transplantation
3. At least one hypo- or dyskinetic segment to demark the implant target area
4. Stable disease condition allowing for an elective left-lateral mini-thoracotomy (for LV applications) or open-chest surgery (for RV applications) for a clinically indicated intervention on the LV (e.g., coronary bypass surgery, valve repair) with concomitant RV dysfunction, diagnosed using the Tricuspid Annular Plane Systolic Excursion (TAPSE) index <16 mm (Rudski et al. 2010).
5. 18-80 years of age
6. Previous implantation of an ICD or CRT-D with event recorder
7. New York Heart Association (NYHA) Class III or IV under optimal medical therapy
8. Willingness and ability to give written informed consent
9. Female subjects of childbearing potential must agree to use acceptable method(s) of contraception for the full study duration.

Exclusion Criteria:

1. Contraindication to immunosuppressive drugs (e.g. known history of unresolved cancer, hepatitis B/C, HIV, HTLV1)
2. Alloimmunisation against EHM implant cells
3. Hypertrophic cardiomyopathy (HCM)
4. Terminal kidney failure (stage 4; GFR <30 ml/min)
5. Terminal liver failure
6. Autoimmune disease
7. History of stroke
8. Reduced life expectancy in the short term due to non-cardiac disease
9. Simultaneous participation in another interventional trial
10. Pregnant or breastfeeding females
11. Known or suspected alcohol and/or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Target heart wall thickness | 12 months
  Target heart wall thickness (HWT) as determined by high resolution echocardiography and/or CINE-mode MRI (17-segment model). Primary efficacy analyses are based on the changes in HWT between baseline and 2 weeks, 1 month, 3 months, 6 months and 12 months after implantation. To test for a time effect a one-way Repeated Measures ANOVA will be performed for the primary endpoint. In case of detecting a time effect this is followed by Dunnett-type pairwise comparisons to baseline using paired t-Tests. Due to the explorative character of the efficacy analysis testing will be performed at a 10% two-sided significance level. Mean differences will be reported along with 90% confidence intervals.
Heart wall thickening fraction | 12 months
  Heart wall thickening fraction (HWTF) as determined by high resolution echocardiography and/or CINE-mode MRI (17-segment model). Primary efficacy analyses are based on the changes in HWTF between baseline and 2 weeks, 1 month, 3 months, 6 months and 12 months after implantation. To test for a time effect a one-way Repeated Measures ANOVA will be performed for the primary endpoint. In case of detecting a time effect this is followed by Dunnett-type pairwise comparisons to baseline using paired t-Tests. Due to the explorative character of the efficacy analysis testing will be performed at a 10% two-sided significance level. Mean differences will be reported along with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Seidler, Prof., Principal Investigator — University Medical Center Goettingen; Wolfram-Hubertus Zimmermann, Prof., Study Director — University Medical Center Goettingen
Locations (3):
- Germany (3):
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - University Medical Center Schleswig-Holstein, Lübeck, Schleswig-Holstein